CLINICAL TRIAL: NCT04002388
Title: Objective Measure of Physical Activity and Sedentary Behavior During Cardiac Rehabilitation: Are Patients Achieving Recommendations/Guidelines
Brief Title: Objective Measure of Physical Activity and Sedentary Behavior During Cardiac Rehabilitation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was withdrawn due to impracticalities in logistics during the COVID-19 pandemic.
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Amanda R. Bonikowske, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 18-009494
Record Dates: First submitted 2019-06-26; First posted 2019-06-28 (Actual); Last update posted 2022-03-07 (Actual); Status verified 2022-02

CONDITIONS: Cardiac Rehab; Physical Activity; Blood Markers
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Activity Monitor Group (Experimental): This arm will receive a FitBit and will be asked to wear this for one year
  Interventions: Behavioral: activity monitor group
- Usual Care Group (Active Comparator): The usual care group will NOT receive a FitBit
  Interventions: Behavioral: usual care group

INTERVENTIONS:
Behavioral: activity monitor group — will receive a FitBit and will be asked to wear this for one year
  Arms: Activity Monitor Group
Behavioral: usual care group — will NOT receive a FitBit
  Arms: Usual Care Group

SUMMARY:
Researchers are trying to assess exercise patterns during and after cardiac rehabilitation participation and to compare changes in blood markers and the microbiome before and after rehabilitation.

DETAILED DESCRIPTION:
Study participation involves a visit to Mayo Clinic at 6 months and 1 year after you begin cardiac rehabilitation. In addition to the standard of care cardiac rehab program, which consists of 36 full sessions, you would be randomized to an activity monitor group or a usual care group.

If randomized to the activity monitor group you will receive a FitBit and will be asked to wear this during cardiac rehabilitation and for one year after you complete the program; complete 4 blood draws (at the start of rehab, at the end of rehab, 6 months after finishing rehab and 1 year after completing rehab) and complete questionnaires about your lifestyle, sleep, mood. The data from the FitBit will be sent to the study team for one year.

If randomized to the usual care group you will complete 4 blood draws (at the start of rehab, at the end of rehab, 6 months after rehab, and 1 year after completing rehab); and complete questionnaires about your lifestyle, sleep, mood.

If you agree to be in the study, you will be asked to wear monitors with capabilities to detect your heart rate or physical activity for up to 1 year. Data will be acquired from the monitors or remote device accounts.

You will also be asked to fill out questionnaires about your current level of physical activity, dietary intake, mood, stress, motivation, and quality of life.

You will have a blood draw.

You will be asked to complete 2 different stool sample tests, saliva tests, and a fingerstick measure for glycosylated hemoglobin; performed at 4 time points.

Information from your medical record will be recorded and used.

ELIGIBILITY:
Inclusion Criteria:

* Adult 18 years and older
* English speaking
* Able to provide consent
* Has a qualifying indication for cardiac rehabilitation (ie. Acute coronary syndrome, myocardial infarction, percutaneous coronary intervention, coronary artery bypass grafting, and stable angina), owns a smart phone and able to download the fitness monitor app (and willing to have their data downloaded from their fitness monitor after completion of cardiac rehab), and able to participate in cardiac rehabilitation.

Exclusion Criteria:

* Does not own a smart phone or is unwilling to download the app or is unable to participate in cardiac rehab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Physical activity measured by Fitbit (steps) | 1 year
  Objective measure of physical activity during cardiac rehabilitation participation and for one year after using a Fitbit and Fitabase.
Amount of time spent sedentary based on activity counts | 1 year
  Objective measure of sedentary time using an accelerometer (activity count levels)
Change in plasma ceramides | 1 year
  Examine the effect of cardiac rehabilitation on plasma ceramide levels

SECONDARY OUTCOMES:
Microbiome changes following an exercise program - Cardiac Rehab | 15 months
  Examine changes in the microbiome and transcriptome following participation in cardiac based on stool, saliva, and biological markers

CONTACTS AND LOCATIONS:
Overall Officials: Amanda R Bonikowske, Principal Investigator — Mayo Clinic

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials